CLINICAL TRIAL: NCT00863200
Title: Identification and Treatment of Depression in Underserved African American and Latino Patients With Cancer
Brief Title: Identification and Treatment of Depression
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0327
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Depression; Cancer; African Americans; Latinos; Hispanics; Interactive voice response; IVR; Behavioral Intervention
MeSH Terms: conditions — Neoplasms; Depression | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telephone Intervention Group
  Interventions: Behavioral: Telephone Intervention; Behavioral: Questionnaires & Interviews
- Standard Care Group
  Interventions: Behavioral: Questionnaires & Interviews

INTERVENTIONS:
Behavioral: Telephone Intervention — Symptom information will be collected using an automated telephone system, approximately 5 minutes per week.
  Other Names: Interactive voice response; IVR
  Groups: Telephone Intervention Group
Behavioral: Questionnaires & Interviews — 3 questionnaires and one-on-one interviews during 3 regularly scheduled clinic visits.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn how well a telephone system works for improving the management of emotional distress, sadness, and/or depression in patients who are being treated for cancer.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups: telephone intervention or standard care. You have an equal chance of being assigned to either group.

No matter which group you are assigned to, you will be asked to tell your doctor and/or nurse about all symptoms you may be experiencing during your regularly scheduled visits. You will also be asked to call your doctor and/or nurse right away when your symptoms are severe. The doctor and/or nurse will give you instructions about calling when your symptoms are severe.

You will receive educational material about emotional distress, sadness, and depression in people who are being treated for cancer. The material also will tell you about community resources that are available for people with cancer.

Feedback Group:

If you are assigned to the feedback group, your symptom information will be collected using a telephone system. You will be asked to rate 13 symptoms, such as sadness, emotional distress, and fatigue, on a scale of 0 to 10 using the touch tone key pad of your telephone. The 0 means that you are not having the symptom at all, and the 10 means that the symptom is as bad as you can imagine.

If you rate either of the 2 symptoms of sadness and/or emotional distress as moderate or severe, then the telephone system will send a message to the research staff and your doctor or nurse right away. Only the symptoms of sadness and emotional distress will be reported right away to the doctor or nurse and the research staff. If you answer moderate to severe to any other questions, it will not be sent right away to the doctor, nurse or study staff. The telephone system usually works very well. But, if for any reason the telephone system is not working, the research staff will report any moderate or severe sadness or distress to your doctor or nurse. Your doctor or nurse also will receive a written summary of your symptom ratings before your next clinic visit.

Standard Care Group:

If you are assigned to the standard care group, your symptom information will not be collected using the telephone system. You will be asked to tell your doctor and/or nurse about all symptoms you may be experiencing.

Telephone System:

For patients in the feedback group, the research staff will teach you how to use a telephone system for measuring your symptoms. The research staff also will ask you to practice using the telephone system. The telephone system will call you 1 time a week for 16 weeks. You will be asked to rate your symptoms and how much the symptoms interfere with your life. You can set up a time to receive the phone calls that works best for you. Rating your symptoms using the telephone system will take about 5 minutes for each call.

If you do not answer the telephone system on the first call, then the system will try to reach you 3 more times. If you do not answer after the fourth try, then the research staff will call you to find out why you could not answer the telephone system. If you prefer, the research staff will change the day or time that the telephone system calls you.

Questionnaires and Interviews:

You will be asked to fill out 3 questionnaires during 3 regularly scheduled clinic visits. These questionnaires ask questions about pain, stress, sadness, quality of life, and other symptoms you may be experiencing. You will also compete an interview at the first and third visit. During the interview, you will be asked questions about your feelings and emotions. The questionnaires and interview will be completed at the following times:

* At the first visit when you enroll in the study, 8-10 weeks after the study begins, and 14-16 weeks after the study begins, you will complete the questionnaires. This will take about 45 minutes.
* At the first visit and 14-16 weeks after the study begins, you will complete a short interview. Completing the interview will take about 15 minutes.

Length of Study:

Your participation in this study will last up to 16 weeks.

This is an investigational study.

Up to 166 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Self-identified as African American or Latino
3. English or Spanish speaking
4. 18 years of age or older
5. Receiving treatment in the medical oncology, genitourinary oncology, or gynecologic oncology clinics at LBJ General Hospital
6. Reports a level of "4" or greater on the MDASI "sadness" and/or "distress" items.

Exclusion Criteria:

1) Not willing to use a telephone to report symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American or Hispanics over 18 years of age being treated for cancer at LBJ General Hospital in Houston.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Learn how well a telephone system works for improving the management of emotional distress, sadness, and/or depression in patients who are being treated for cancer. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Tito Mendoza, BS,MED,MS,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- LBJ General Hospital, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org